CLINICAL TRIAL: NCT01013701
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Single Center Study to Compare the Effects of Fluticasone Furoate Nasal Spray vs Placebo in Patients With Nasal Polypoid Disease
Brief Title: Compare the Effects of Fluticasone Furoate Nasal Spray vs Placebo in Patients With Nasal Polypoid Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated based on mutual agreement between PI and sponsor (Glaxo Smith Kline)
Sponsor: Johns Hopkins University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NA_00029405
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Results first posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-08

CONDITIONS: Patients With Nasal Polyps
Keywords: nasal polyps; nasal steroid; fluticasone furoate
MeSH Terms: conditions — Nasal Polyps | interventions — fluticasone furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluticasone Furoate (Active Comparator): nasal steroid
  Interventions: Drug: fluticasone furoate
- Placebo (Placebo Comparator): nasal spray vehicle without drug
  Interventions: Other: placebo

INTERVENTIONS:
Drug: fluticasone furoate — nasal steroid spray
  Arms: Fluticasone Furoate
Other: placebo — nasal steroid vehicle without drug
  Arms: Placebo

SUMMARY:
Fluticasone furoate is being studied to determine whether treatment with a topical nasal steroid, in patients with existing nasal polyps , can not only improve symptoms but also suppress the recurrence of clinically significant nasal polyp obstruction and prevent surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 18-70 years of age, in general good health.
2. Current evidence of nasal polyps on physical exam. 3) Able to understand the protocol and comply with instructions. 4) Have a negative urine pregnancy test in women of childbearing potential. 5) Women of childbearing potential must be on an acceptable method of birth control or willing to remain abstinent through the duration of the study.

Exclusion Criteria:

1. Are pregnant and/or breast-feeding.
2. History of alcohol or drug abuse in the past year.
3. Signs and symptoms suggestive of fulminant bacterial sinusitis (fever >101 F, persistent severe unilateral facial or tooth pain, facial swelling).
4. Allergies to nasal corticosteroids
5. .Other chronic significant medical illnesses 6) Maintenance oral prednisone therapy for other chronic medical conditions.

   -

   -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2010-07-29 (Actual); Study Completion 2010-07-29 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The PI has left the institution and neither he, nor the data if any, is available. All information provided has been obtained from the Johns Hopkins University School of Medicine Institutional Review Board and was only available as one arm.
Groups:
- All Participants: nasal steroid fluticasone furoate: nasal steroid spray
  OR
  nasal spray vehicle without drug placebo: nasal steroid vehicle without drug
Period: Overall Study
Arm/Group | All Participants
Started | 7
Completed | 0
Not Completed | 7
Not completed — study prematurely terminated | 7

BASELINE CHARACTERISTICS:
Population: The PI has left the institution and neither he, nor the data if any, is available. All information provided has been obtained from the Johns Hopkins University School of Medicine Institutional Review Board and was only available as one arm.
Arm/Group | All Participants
Number analyzed (Participants) | 7
Age, Customized [Count of Participants; unit: Participants]
  >=18, <=70, years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Effect of Once Daily Nasal Steroid Therapy With Fluticasone Furoate Nasal Spray (110 mcg/Day) in Suppressing Nasal Polyp-induced Symptoms Over the Course of 16 Weeks in Patients Presenting to the Clinic With Active Nasal Polypoid Disease.
Time Frame: 18 weeks
Population: The PI has left the institution and neither he, nor the data if any, is available. All information provided has been obtained from the Johns Hopkins University School of Medicine Institutional Review Board.
Groups:
- Nasal Steroid: nasal steroid fluticasone furoate: nasal steroid spray
- Placebo: nasal spray vehicle without drug placebo: nasal steroid vehicle without drug
Arm/Group | Nasal Steroid | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: To Evaluate the Efficacy and Safety of Once Daily Nasal Steroid Therapy With Fluticasone Furoate Nasal Spray in Suppressing the Signs of Recurrence of Nasal Polyps Over the Course of 16 Weeks.
Time Frame: 18 weeks
Population: No data was collected/is available for the study as it was terminated prematurely and the PI has since left the institution.
Arm/Group | Nasal Steroid | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: No data was collected/is available for the study as it was terminated prematurely and the PI has since left the institution. The information in Adverse events is presenter per arm, as the arm assignment, if any, is unknown.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes